CLINICAL TRIAL: NCT05101681
Title: Diagnostic Accuracy of Teledentistry Versus Direct Oral Examination of Elderly in Aged-Care Homes: A Pilot Cross-Sectional Study
Brief Title: Accuracy of Teledentistry Versus Direct Oral Examination for Elderly in Aged-Care Homes: A Pilot Cross-Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatollah Nagy Sharkawy Ali Nada, Dr., Cairo University
Other Study IDs: Teledentistry for Elderly
Record Dates: First submitted 2021-10-29; First posted 2021-11-01 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Oral Screening for Elderly in Aged Care Homes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Teledentistry — Teledentistry using mobile photographs

SUMMARY:
The residents will receive oral health education, then three examiners ( licensed dentists ) will perform the direct oral examination of the participants. During the same visit, a dental student will take the intraoral photographs in the aged care home.

Later, three different blinded examiners (licensed dentists) will assess the intraoral photographs of the same group of participants. The participant's dentition will be examined using the scores developed by the World Health Organization (WHO) for oral health surveys. Also, the examiners will perform a visual inspection of the oral mucosa for any signs of oral potentially malignant disorders (OPMD), as the mortality of high-risk populations is proven to be reduced by visual oral cancer screening.

Finally, the residents who require treatment will be referred to Kasr EL Ainy dental hospital to receive dental treatments.

DETAILED DESCRIPTION:
The residents will receive oral health education, by three examiners ( licensed dentists ) with a t least 5 years experience. Then the same examiner will perform the direct oral examination of the participants. They will fill the dentition status, denture status, oral lesions and intervention urgency section of the World Health Organization (WHO) form 2013 version.

During the same visit, a dental student will take the intraoral photographs in the aged care home. The photographs will include 5 views (upper occlusal, lower occlusal , frontal, right lateral and left lateral).

The photographs will be uploaded on one drive and later, three different blinded examiners (licensed dentists) will assess the intraoral photographs of the same group of participants. The participant's dentition will be examined using the scores developed by the World Health Organization (WHO) for oral health surveys. Also, the examiners will perform a visual inspection of the oral mucosa for any signs of oral potentially malignant disorders (OPMD), as the mortality of high-risk populations is proven to be reduced by visual oral cancer screening.

Finally, the residents who require treatment will be referred to Kasr EL Ainy dental hospital to receive dental treatments.

ELIGIBILITY:
Inclusion Criteria:

* Elderly living in aged care homes in Egypt
* Have the ability to communicate with the examiner
* Have the ability to give consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants are elderly living in aged care homes in Egypt who must be able to communicate with the examiner and must be able to give consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dentition status | January- December 2023
  Feasibility of tele dentistry mobile photographic method to assess the dentition status of the elderly living in elderly homes will be measured by comparing the tele dentistry method with the direct oral examination .The scores of the World Health Organization (WHO) assessment forms of oral health will be used with the crowns.
  Also, the dentures section will be used to record the presence or absence of partial or complete dentures in both jaws.

SECONDARY OUTCOMES:
Oral Mucosal lesions | January- December 2023
  Signs for Oral potentially malignant disorders OPMD visible in the photographic views and direct examination will be recorded in the section of the oral mucosal lesions in the assessment form .This will be performed by the direct examiners and the tele dentistry examiners to compare both methods of examination.

OTHER OUTCOMES:
Intervention Urgency | January- December 2023
  The intervention urgency section in the World Health Organization (WHO) form will be used for the assessment of the triaging of the elderly.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Dar El Sahwa Elderly Home, Giza
  - Khadmat El Mogtamaa Elderly Home, Giza